CLINICAL TRIAL: NCT01743794
Title: Efficacy of Continuous Wound Infusion in Major Lumbar and Thoracic Spine Surgery : A Randomised, Double-blinded, Placebo-controlled Study
Brief Title: Continuous Wound Infusion in Lumbar or Thoracic Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1008
Record Dates: First submitted 2012-05-09; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Lumbar Spine Surgery; Thoracic Spine Surgery
MeSH Terms: interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ropivacaine 0.2%, wound infusion (Experimental)
  Interventions: Drug: Ropivacaine
- saline solution 0.9%, wound infusion (Placebo Comparator)
  Interventions: Drug: Saline solution 0.9%

INTERVENTIONS:
Drug: Ropivacaine — wound infusion, 0.2%, bolus 10mL followed by 8 mL/h infusion
  Arms: ropivacaine 0.2%, wound infusion
Drug: Saline solution 0.9% — wound infusion, 0.9%, bolus 10mL followed by 8 mL/h
  Arms: saline solution 0.9%, wound infusion

SUMMARY:
Introduction : Spine surgery is responsible for intense postoperative pain that can be treated by an analgesia multimodal approach (IV analgesic infusion and local anesthesia). Continuous wound infiltration is an efficient and simple technique with few adverse effects yet very few studies have investigated its potential use in spine surgery. Our randomised, controlled, double-blinded trial aims to evaluate efficacy of continuous wound infiltration after major spine surgery.

Methods : After written consent is obtained, the surgeon inserts, at the end of surgery, a multiholes catheter under muscular layers. Patients are randomised in two groups : The "treated group" receives ropivacaine 0.2% infusion (bolus of 10 milliliters (mL) followed by 8 mL/h continuous infusion during 48 hours) and the "control group" receives saline solution (0.9%). In addition, all patients receive patient-controlled intra-venous morphine analgesia. The investigators hypothesize that the "treated group" will consume morphine less than the "control group".

ELIGIBILITY:
Inclusion Criteria:

* adults
* > 18 years
* Physical status score I, II or III (American Society of Anesthesiologists)
* lumbar or thoracic spine surgery with arthrodesis through posterior only approach
* signed informed consent
* beneficiary of social security

Exclusion Criteria:

* vulnerable persons according to law
* scoliosis surgery
* local anesthetic allergia
* contraindication to ketamine, acetaminophene, nefopam, non steroidal anti inflammatory, ropivacaine, morphine, droperidol
* long term anti platelet aggregants
* inability to comply to protocol requirements
* psychiatric disorders or cognitive disabilities
* chronic pain or long term opioids consumption
* diabetes
* obesity (BMI > 30)
* pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
morphine consumption | 48 hours after surgery

SECONDARY OUTCOMES:
number of patients in need of morphine in post surgery monitoring room | 1 hour after surgery
morphine consumption in post surgery monitoring room | 1 hour post surgery
consumption of morphine | 72 hours after surgery
global self appreciation of pain management | at 72 hours
Time required for post surgery functional recovery | participants will be followed for the duration of hospital stay, an expected average of 3 weeks
Adverse effects of morphine | 72 hours after surgery
hospitalization delay | participants will be followed for the duration of hospital stay, an expected average of 3 weeks
asked bolus divided by delivered bolus | until 72 hours after surgery
Score for pain intensity | until 72 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Departement of Anesthesia and Intensive Care, Grenoble, Auvergne-Rhône-Alpes, France

REFERENCES:
- [Derived] Greze J, Vighetti A, Incagnoli P, Quesada JL, Albaladejo P, Palombi O, Tonetti J, Bosson JL, Payen JF. Does continuous wound infiltration enhance baseline intravenous multimodal analgesia after posterior spinal fusion surgery? A randomized, double-blinded, placebo-controlled study. Eur Spine J. 2017 Mar;26(3):832-839. doi: 10.1007/s00586-016-4428-1. Epub 2016 Feb 10. PMID 26865083